CLINICAL TRIAL: NCT05502835
Title: Pulse Pressure Variation Based Intraoperative Fluid Management Versus Traditional Fluid Management for Colonic Cancer Patients Undergoing Mass Resection and Anastomosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, Assistant Professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00006379 GUT OEDEMA
Record Dates: First submitted 2022-08-02; First posted 2022-08-16 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Intraoperative Fluid Volume; Hemodynamics; Serum Lactate; Intestinal Edema; Length of the Hospital Stay; First Time to Gastrointestinal Motion; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional fluid management group (Experimental): patients will do elective open colonic mass resection and anastomosis will receive Infusion of 6 ml/kg/hr. Ringer's solution.
  Interventions: Other: conventional fluid management
- ppv group (Active Comparator): patients will do elective open colonic mass resection and anastomosis. Infusion of 2 ml/kg/hr. Ringer's solution guided by pulse pressure variation.
  Interventions: Device: pulse pressure variation

INTERVENTIONS:
Device: pulse pressure variation — Infusion of 2 ml/kg/hr. Ringer's solution guided by pulse pressure variation.
  Arms: ppv group
Other: conventional fluid management — Infusion of 6 ml/kg/hr. Ringer's solution.
  Arms: conventional fluid management group

SUMMARY:
pulse pressure variation based intraoperative fluid therapy versus traditional fluid therapy for colonic cancer patients undergoing mass resection and anastomosis for maintaining adequate hydration without complications.

DETAILED DESCRIPTION:
All Patients will be assigned randomly by using computerized program to one of the two equal groups. Patients will be (forty five patients per group):

Group A ;( control group) Forty five patients will do elective open colonic mass resection and anastomosis. Infusion of 6 ml/kg/hr. Ringer's solution.

Group B; Forty five patients will do elective open colonic mass resection and anastomosis. Infusion of 2 ml/kg/hr. Ringer's solution guided by pulse pressure variation.

Intraoperative fluid volume, hemodynamics, serum lactate and intestinal edema will be measured after induction of anesthesia and every hour till the end of the operation, length of the hospital stay, first time to gastrointestinal motion and postoperative complications are recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status (ASA-PS) I and II Patients.
* Patients scheduled for elective open colonic mass resection and anastomosis.

Exclusion Criteria:

* Serious cardiac arrhythmia.
* Peripheral artery disease.
* An ejection fraction below 30%.
* A pulmonary pathology.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — participant eligibility is based on self-representation of gender identity
Enrollment: 90 (Actual)
Dates: Start 2022-08-20 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Intraoperative fluid volume | calculated immediately after surgery

SECONDARY OUTCOMES:
intraoperative blood pressure | every ten minutes till the end of the surgery
lactate level | every hour till the end of the surgery
POSTOPERATIVE COMPLICATIONS | till one week after surgery
intestinal oedema | intraoperatively after tumor resection

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No